CLINICAL TRIAL: NCT04137523
Title: INVESTIGATING eNAMPT ROLE IN ACQUISITION OF EPITHELIAL TO MESENCHYMAL TRANSITION-LIKE FEATURES IN MULTIPLE MYELOMA
Brief Title: Investigate eNAMPT in Multiple Myeloma Biology and Establish Its Role in Disease Progression
Status: Completed | Type: Observational
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Dr. Alessandra Larocca, Principal Investigator, University of Turin, Italy
Other Study IDs: eNAMPT
Record Dates: First submitted 2019-10-21; First posted 2019-10-24 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Multiple Myeloma
Keywords: potential marker; cytokine/adipokine; multiple myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Based on our previous observations, here the investigator plans to further investigate eNAMPT in MM biology and to establish its role in disease progression where EMT acquisition represents an hallmark of cancers. Results deriving from proposal would hopefully identify novel biological vulnerabilities of such malignancy and an innovative biomarker for disease progression monitoring as well.

DETAILED DESCRIPTION:
Background and preliminary data:

Multiple myeloma (MM) is characterized by a clonal expansion of malignant plasma cells in the bone marrow (BM) with a continuous spread of tumour cells in and out of BM. A continuous interaction between BM stromal cells (BMSCs) and MM cells supports proliferation, survival, migration, and drug resistance of tumor cells. Indeed, BMSCs by both cytokines production and cell-cell interactions, control the ability of MM cells to enter into bloodstream, leading to homing or extravasation of clonal cells into distant tissues, which in turn results in new BM niches formation.

The epithelial-to-mesenchymal transition (EMT) is a biological phenomenon by which epithelial cells can switch into a mesenchymal phenotype through the disruption of cell-cell adhesion and cellular polarity, remodeling of cytoskeleton and changing cell-matrix adhesion. Overall, these events lead to improved migratory and invasive properties of affected cells. Remarkably, EMT occurs physiologically during normal embryonic development and tissue regeneration but, in cancer cell, it has been associated with tumor aggressiveness features including invasion, metastasis, stemness and drug-resistance. EMT is commonly observed in solid tumors but it has been recently described also in MM. In such a context, studies have shown that BM niches-associated hypoxia produces MM cells egress and dissemination through acquisition of EMT-like features which in turn, by increasing CXCR4 expression, produces extra-medullary disease (EMD) development.

Alterations in cell metabolism have emerged as one of the hallmarks of cancer that could be possibly targeted by novel therapeutic approaches. Among these alterations, biosynthesis of nicotinamide adenine dinucleotide (NAD+) is emerging as novel therapeutic target in tumours. Nicotinamide phosphorybosyltransferase (NAMPT), the rate-limiting enzyme for NAD+ production from nicotinamide (NAM) in mammalian cells, is frequently up-regulated in cancers, including MM, and its relevance as potential therapeutic target has been widely explored by our group. However, beside its intracellular activity as key metabolic enzyme, NAMPT is also present in the extracellular milieu where it exerts cytokine/adipokine-like actions as eNAMPT. Although mechanisms underlying eNAMPT secretion still remain to be elucidated, it is commonly accepted that there is positive correlation between eNAMPT secretion and intracellular NAMPT levels. Recent evidences show that eNAMPT plasma levels are significantly higher in cancer patients in comparison with healthy donors in several hematologic and solid neoplasms. In this context, eNAMPT was found to exert pro-tumorigenic effects such as promoting cancer cell proliferation and colonies formation, conferring resistance to apoptosis and shaping of tumour microenviroment, by promoting neo-angiogenesis and affecting immune response.

The Investigators recently demonstrated the pivotal role played by eNAMPT in the acquisition of EMT in human breast cancer cells. In detail, NAMPT overexpression promotes acquisition of fibroblast-like morphology of cancer cells by reducing E-cadherin expression in association with N-cadherin, Vimentin and ZEB1 upregulation. Importantly, NAMPT-induced EMT is not associated with NAMPT enzymatic activity and neither with its product levels nicotinamide mononucleotide (NMN). On the contrary, EMT seems to be mediated by eNAMPT through its ability to activate TGFβ signaling pathway via increased TGFβ1 production.

Based on our previous observations, here the investigators plan to further investigate eNAMPT in MM biology and to establish its role in disease progression where EMT acquisition represents an hallmark of cancers. Results deriving from proposal would hopefully identify novel biological vulnerabilities of such malignancy and an innovative biomarker for disease progression monitoring as well.

The investigators have preliminary measured eNAMPT serum levels in PB samples of Newly Diagnosed Multiple Myeloma (NDMM) (n= 20) patients and healthy donors (HDs; n=6). Interestingly, eNAPMT levels were found to be significantly higher in tumors than controls, pointing to a relevant role of this cytokine in MM biology. These data provide the rationale for further investigations of eNAMPT role in MM.

Sample collection:

Retrospective samples of MM patients will be derived from two different databases (UNITO and UNIGE) and combined into a new specific database dedicated to this project to cover the different stages of disease that will be analyzed.

UNITO will coordinate and perform the selection of the samples that will be included. UNITO will be able to provide the required number of samples for this study. Ultimately, an independent, representative set of 100 MM patient samples will be selected from previous clinical trials that have been conducted over the past 5 years.

In general, the samples will meet the following parameters:

* Male and female patients over 18 years of age;
* PB-derived serum samples collected in different disease phases (MGUS, SMM, NDMM and RRMM MM patients)
* Sufficient CD138+ cells or RNA from CD138+ cells are available;
* ≥ 2 years median survival data and treatment data is available (progression free and overall survival);
* Bone marrow sample acquired prior to the initiation of the therapy of interest;
* Patients have consented for use of their sample for research purposes.

A feasibility assessment and power analysis of the available samples and clinical data will be performed for each of the respective available clinical trials from which the samples will originate. This assessment is performed in order to decide upon, select, and build, a dataset that provides scientifically and statistically sound evidence for treatment effectiveness prediction. The selected treatment regimens (combinations of medication) that will be analyzed cover the complete spectrum of MM treatment classes, including proteasome inhibitors, immunomodulatory drugs (IMiDs), alkylating agents, HDAC inhibitors and monoclonal antibodies. Patient samples will be derived from controlled clinical trials, and will be selected from different treatment groups, containing patients that received the same treatment regimens, based on one of the following drugs or combinations: Bortezomib (proteasome inhibitor), Carfilzomib (proteasome inhibitor), Thalidomide (IMiD), Lenalidomide (IMiD), Pomalidomide (IMiD), Melphalan (alkylating agent), Panabinostat (HDAC inhibitor), and Daratumumab (monoclonal antibody).

Sample size estimations are based on previous experiences of being able to significantly determine survival differences between positive and negative cases for a certain treatment for a sufficiently large group. Given an effect size of at least 3 and an incidence of the subtype of 20%, a group size of 100 cases will be sufficient to significantly determine the predictive value of the subtype. (a smaller effect size and a smaller incidence would likely not be clinically relevant).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients over 18 years of age;
* PB-derived serum samples collected in different disease phases (MGUS, SMM, NDMM and RRMM MM patients)
* Sufficient CD138+ cells or RNA from CD138+ cells are available;
* ≥ 2 years median survival data and treatment data is available (progression free and overall survival);
* Bone marrow sample acquired prior to the initiation of the therapy of interest;
* Patients have consented for use of their sample for research purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 MM patient samples will be selected from previous clinical trials that have been conducted over the past 5 years.
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
To strengthen preliminary data | 2 years
  To strengthen preliminary data and to investigate the correlation between eNAMPT levels in BM and peripheral blood (PB) compartments by assessing its concentration in paired samples collected from a larger cohort of NDMM patients, using also more HDs as control.
Potential marker of PD | 2 years
  To disclose eNAMPT relevance as potential marker of disease progression by comparing eNAMPT plasmatic levels from samples collected in different phases of disease (MGUS, Smoldering Multiple Myeloma -SMM-, NDMM, relapsed/refractory MM) and by their correlation with available clinical data.
Analysis both MM cells and MM-BMSC compartment. | 2 years
  To investigate cellular source of eNAMPT production in MM by analyzing both MM cells (Established Human Myeloma Cell Lines, HMCLs and primary CD138+ cells) and MM-BMSC compartment.
To investigate eNAMPT role | 2 years
  To investigate eNAMPT role in EMT features acquisition of HMCLs (with known molecular features such as karyotype status, mutations, drug-resistance phenotype etc.) and to define the underlying molecular mechanisms.
To determine the effects | 2 years
  To determine the effects of previously identified neutralizing αeNAMPT antibody (Ab) (13) on MM cells both in vitro and in an in vivo MM-xenografted mouse model.

CONTACTS AND LOCATIONS:
Locations (1):
- Aou Citta' Della Salute E Della Scienza Di Torino, Torino, TO, Italy

IPD SHARING:
Plan to Share IPD: Undecided